CLINICAL TRIAL: NCT02457598
Title: A Phase 1b Dose Escalation and Dose Expansion Study of Tirabrutinib (ONO/GS-4059) in Combination With Other Targeted Anti-cancer Therapies in Subjects With B-cell Malignancies
Brief Title: Dose Escalation and Dose Expansion Study of Tirabrutinib in Combination With Other Targeted Anti-cancer Therapies in Adults With B-cell Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The goal of the study was to improve tolerability while maintaining or increasing efficacy. The results of this study showed no efficacy advantage although the combinations were well tolerated.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-401-1757; 2015-000834-30 (EudraCT Number)
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Results first posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: B-cell Malignancies
MeSH Terms: interventions — tirabrutinib; idelalisib; 6-(1H-indazol-6-yl)-N-(4-morpholinophenyl)imidazo(1,2-a)pyrazin-8-amine; obinutuzumab

STUDY DESIGN:
Intervention Model Description: Enrollment and treatment were parallel in different combinations used in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (17):
- Combination I (Tirabrutinib 20 mg QD+ Idelalisib 50 mg BID) (Experimental): Participants will receive tirabrutinib 20 mg tablet once daily (QD) for up to 209 weeks and idelalisib 50 mg tablet twice daily (BID) orally for up to 120 weeks. Both drugs will be administered for 28-day cycles.
  Interventions: Drug: Tirabrutinib; Drug: Idelalisib
- Combination I (Tirabrutinib 40 mg QD+ Idelalisib 50 mg BID) (Experimental): Participants will receive tirabrutinib 40 mg tablet QD for up to 251 weeks and idelalisib 50 mg tablet BID orally, for up to 245 weeks. Both drugs will be administered for 28-day cycles.
  Interventions: Drug: Tirabrutinib; Drug: Idelalisib
- Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID) (Experimental): Participants will receive tirabrutinib 80 mg tablet QD for up to 212 weeks and idelalisib 50 mg tablet BID orally, for up to 26 weeks. Both drugs will be administered for 28-day cycles.
  Interventions: Drug: Tirabrutinib; Drug: Idelalisib
- Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD) (Experimental): Participants will receive tirabrutinib 80 mg tablet QD for up to 227 weeks and idelalisib 100 mg tablet QD orally, for up to 227 weeks. Both drugs will be administered for 28-day cycles.
  Interventions: Drug: Tirabrutinib; Drug: Idelalisib
- Combination I (Tirabrutinib 160 mg QD+ Idelalisib 100 mg QD) (Experimental): Participants will receive tirabrutinib 160 mg tablet QD for up to 151 weeks and idelalisib 100 mg tablet QD orally, for up to 151 weeks. Both drugs will be administered for 28-day cycles.
  Interventions: Drug: Tirabrutinib; Drug: Idelalisib
- Combination I (Tirabrutinib 20 mg BID+ Idelalisib 50 mg BID) (Experimental): Participants will receive tirabrutinib 20 mg tablet BID for up to 207 weeks and idelalisib 50 mg tablet BID orally, for up to 207 weeks. Both drugs will be administered for 28-day cycles.
  Interventions: Drug: Tirabrutinib; Drug: Idelalisib
- Combination II (Tirabrutinib 40 mg QD+ Entospletinib 200 mg QD) (Experimental): Participants will receive tirabrutinib 40 mg tablet QD for up to 250 weeks and entospletinib 200 mg tablet QD orally, for up to 250 weeks. Both drugs will be administered for 28-day cycles.
  Interventions: Drug: Tirabrutinib; Drug: Entospletinib
- Combination II (Tirabrutinib 80 mg QD+ Entospletinib 200 mg QD) (Experimental): Participants will receive tirabrutinib 80 mg tablet QD for up to 234 weeks and entospletinib 200 mg tablet QD orally, for up to 220 weeks. Both drugs will be administered for 28-day cycles.
  Interventions: Drug: Tirabrutinib; Drug: Entospletinib
- Combination II (Tirabrutinib 150 mg QD+ Entospletinib 200 mg QD) (Experimental): Participants will receive tirabrutinib 150 mg tablet QD for up to 103 weeks and entospletinib 200 mg tablet QD orally, for up to 88 weeks. Both drugs will be administered for 28-day cycles.
  Interventions: Drug: Tirabrutinib; Drug: Entospletinib
- Combination II (Tirabrutinib 40 mg QD+ Entospletinib 400 mg QD) (Experimental): Participants will receive tirabrutinib 40 mg tablet QD for up to 119 weeks and entospletinib 400 mg tablet QD orally, for up to 119 weeks. Both drugs will be administered for 28-day cycles.
  Interventions: Drug: Tirabrutinib; Drug: Entospletinib
- Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD) (Experimental): Participants will receive tirabrutinib 80 mg tablet QD for up to 232 weeks and entospletinib 400 mg tablet QD orally, for up to 229 weeks. Both drugs will be administered for 28-day cycles.
  Interventions: Drug: Tirabrutinib; Drug: Entospletinib
- Combination II (Tirabrutinib 160 mg QD+ Entospletinib 400 mg QD) (Experimental): Participants will receive tirabrutinib 160 mg tablet QD for up to 44 weeks and entospletinib 400 mg tablet QD orally, for up to 44 weeks. Both drugs will be administered for 28-day cycles.
  Interventions: Drug: Tirabrutinib; Drug: Entospletinib
- Combination III (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD+ obinutuzumab 1000 mg) (Experimental): Participants will receive tirabrutinib 80 mg tablet QD for up to 199 weeks; Idelalisib 100 mg tablet QD orally for up to 199 weeks, and single dose of obinutuzumab 1000 mg intravenously (IV) for up to 22 weeks. Both drugs will be administered for 28-day cycles.
  Interventions: Drug: Tirabrutinib; Drug: Idelalisib; Drug: Obinutuzumab
- Combination IV (Tirabrutinib 80 mg QD+ entospletinib 400 mg QD+ obinutuzumab 1000 mg) (Experimental): Participants will receive tirabrutinib 80 mg tablet QD for up to 196 weeks; entospletinib 400 mg tablet QD orally for up to 196 weeks and single dose of obinutuzumab 1000 mg IV for up to 22 weeks. Both drugs will be administered for 28-day cycles.
  Interventions: Drug: Tirabrutinib; Drug: Entospletinib; Drug: Obinutuzumab
- Group V Single Agent Tirabrutinib (Experimental): Participants will receive tirabrutinib 80 mg tablet QD orally, for each 28-day cycle up to 194 weeks.
  Interventions: Drug: Tirabrutinib
- Group VI Single Agent Tirabrutinib: CLL (Experimental): Participants with CLL who received tirabrutinib in this or a previous tirabrutinib study will continue to receive tirabrutinib at the original dose (between the range of 40 - 400 mg), tablet QD, for each 28-day cycle up to 441 weeks. Participants will be monitored for the long-term safety of tirabrutinib in this group.
  Interventions: Drug: Tirabrutinib
- Group VI Single Agent Tirabrutinib: NHL (Experimental): Participants with NHL who received tirabrutinib in this or a previous tirabrutinib study will continue to receive tirabrutinib at the original dose (between the range of 60 - 480 mg), tablet QD, for each 28-day cycle up to 441 weeks. Participants will be monitored for the long-term safety of tirabrutinib in this group.
  Interventions: Drug: Tirabrutinib

INTERVENTIONS:
Drug: Tirabrutinib — Capsules or tablets administered orally
  Other Names: ONO/GS-4059
Drug: Idelalisib — Tablets administered orally twice daily
  Other Names: Zydelig®; GS-1101; CAL-101
  Arms: Combination I (Tirabrutinib 160 mg QD+ Idelalisib 100 mg QD); Combination I (Tirabrutinib 20 mg BID+ Idelalisib 50 mg BID); Combination I (Tirabrutinib 20 mg QD+ Idelalisib 50 mg BID); Combination I (Tirabrutinib 40 mg QD+ Idelalisib 50 mg BID); Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD); Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID); Combination III (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD+ obinutuzumab 1000 mg)
Drug: Entospletinib — Tablets administered orally
  Other Names: GS-9973
  Arms: Combination II (Tirabrutinib 150 mg QD+ Entospletinib 200 mg QD); Combination II (Tirabrutinib 160 mg QD+ Entospletinib 400 mg QD); Combination II (Tirabrutinib 40 mg QD+ Entospletinib 200 mg QD); Combination II (Tirabrutinib 40 mg QD+ Entospletinib 400 mg QD); Combination II (Tirabrutinib 80 mg QD+ Entospletinib 200 mg QD); Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD); Combination IV (Tirabrutinib 80 mg QD+ entospletinib 400 mg QD+ obinutuzumab 1000 mg)
Drug: Obinutuzumab — Administered intravenously
  Arms: Combination III (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD+ obinutuzumab 1000 mg); Combination IV (Tirabrutinib 80 mg QD+ entospletinib 400 mg QD+ obinutuzumab 1000 mg)

SUMMARY:
The primary objectives of this study are to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary efficacy of tirabrutinib (ONO/GS-4059) in combination with other targeted anti-cancer therapies and to evaluate the long-term safety of tirabrutinib as a monotherapy and in combination with other targeted anti-cancer therapies in adults with relapsed or refractory B-cell lymphoproliferative malignancies.

This study consists of three parts: Dose Escalation, Dose Expansion, and Long-term Safety Monitoring. During the Dose Escalation phase, participants will be sequentially enrolled in a standard 3 + 3 dose escalation study design, to receive oral tirabrutinib combined with idelalisib entospletinib +/- obinutuzumab. The Dose Expansion Phase will enroll additional participants with a single B-cell lymphoproliferative malignancy disease type to further evaluate efficacy, safety, tolerability, PK, and pharmacodynamics. The Long-term Safety Monitoring phase will evaluate the long-term safety of tirabrutinib both as a monotherapy and in combination with other anti-cancer therapies. As of Amendment 9, all participants currently on the study who have no clinical evidence of disease progression will transition into long-term safety monitoring. Participants from the ongoing Study GS-US-401-1787 and participants who came off Study GS-US-401-1757 and Study GS-US-401-1787 but continued to receive treatment via named patient use (or individual expanded use) will be enrolled into the long-term safety monitoring group (Group VI). Participants enrolled in Group VI will continue the same treatment regimen in Study GS-US-401-1787 or named patient use (or individual expanded use). As of Protocol Amendment 8, the maximum treatment duration for any participant is an additional 6 years from the date of this amendment (ie. until November 2025). As of Amendment 9, entospletinib will be provided until 31 December 2020 to participants who are currently receiving entospletinib. Participants treated with entospletinib as part of a combination regimen with tirabrutinib will stop receiving entospletinib by 31 December 2020 but may continue to be treated with tirabrutinib monotherapy. Idelalisib will be provided as 50 mg tablets until 31 December 2020 and 100 mg tablets until study completion. Participants assigned to the 50 mg tablet will be given the option, at the investigator's discretion, to switch to 100 mg once daily idelalisib dose.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of follicular lymphoma (FL), marginal zone lymphoma (MZL), small lymphocytic lymphoma (SLL), chronic lymphocytic leukemia (CLL) (meeting International Workshop on Chronic Lymphocytic Leukemia (IWCLL) Criteria 2008), mantle cell lymphoma (MCL), Waldenstrom's macroglobulinemia (WM), or non-germinal center B-cell lymphoma (GCB) diffuse large B-cell lymphoma (DLBCL) as documented by medical records on World Health Organization (WHO) criteria
* Prior treatment for FL, MZL, SLL, MCL, WM with ≥ 2 or for CLL or non-GCB DLBCL ≥ 1 chemotherapy-based or immunotherapy-based regimen, and not transplant eligible and have had either progressive disease (PD) or no response to previous treatment
* For diseases other than Waldenstrom's macroglobulinemia (WM), presence of radiographically measurable presence of ≥ 1 lesion that measures ≥ 2.0 cm in the longest dimension (LD) and ≥ 1.0 cm in the longest perpendicular dimension (LPD)
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Platelets ≥ 50 x 10^9/L; Hb ≥ 8.0 g/dL; absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L
* Without transfusion and growth factors within 7 days
* Aspartate transaminase/alanine transaminase (AST/ALT) ≤ 2.5 x upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 x ULN
* Creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 60 mL/min
* Not pregnant
* Willingness and ability to comply with protocol-specified Pneumocystis jirovecii pneumonia (PJP) prophylaxis
* Long-term Safety Monitoring group only (Group VI):

  * Currently enrolled in Study GS-US-401-1787 or previously enrolled in Study GS-US-401-1757 or Study GS-US-401-1787 and currently receiving continued treatment via named patient use
  * Continuing to benefit from the current treatment regimen in the opinion of the investigator/treating physician

Key Exclusion Criteria:

* Hepatitis B surface antigen (HBsAG) positive or hepatitis B core antibody positive
* Hepatitis C virus (HCV) antibody positive
* History of long QT syndrome or whose corrected QT(QTc) interval measured (Fridericia method) at screening is prolonged (>450 ms)
* Long-term Safety Monitoring group only (Group VI):

  * Evidence of clinical or radiological disease progression

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2015-06-16 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (15):
- United States (3):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Indiana University Health Goshen Center for Cancer Care, Goshen, Indiana
  - Oregon Health and Science University, Portland, Oregon
- France (5):
  - CHRU de Lille, Hopital Claude Huriez, Lille
  - Hopital Saint Eloi, Montpellier
  - Chu Haut Leveque, Pessac
  - Centre Hospitalier de Lyon Sud, Pierre-Bénite
  - Institut Universitaire du Cancer-Oncopole I.U.C.T-O, Toulouse
- United Kingdom (7):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Cardiff and Vale Health Board, Clinical Research Facility, Cardiff
  - Leeds Teaching Hosptials NHS Trust, Dept of Haematology, Leeds
  - University Hospitals of Leicester NHS Trust, Leicester
  - The Christie NHS Foundation Trust, Manchester
  - Plymouth Hospitals NHS Trust, Plymouth
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Danilov AV, Herbaux C, Walter HS, Hillmen P, Rule SA, Kio EA, Karlin L, Dyer MJS, Mitra SS, Yi PC, Humeniuk R, Huang X, Zhou Z, Bhargava P, Jurgensmeier JM, Fegan CD. Phase Ib Study of Tirabrutinib in Combination with Idelalisib or Entospletinib in Previously Treated Chronic Lymphocytic Leukemia. Clin Cancer Res. 2020 Jun 15;26(12):2810-2818. doi: 10.1158/1078-0432.CCR-19-3504. Epub 2020 Mar 10. PMID 32156743
- [Background] Morschhauser F, Dyer MJS, Walter HS, Danilov AV, Ysebaert L, Hodson DJ, Fegan C, Rule SA, Radford J, Cartron G, Bouabdallah K, Davies AJ, Spurgeon S, Rajakumaraswamy N, Li B, Humeniuk R, Huang X, Bhargava P, Jurgensmeier JM, Salles G. Phase 1b study of tirabrutinib in combination with idelalisib or entospletinib in previously treated B-cell lymphoma. Leukemia. 2021 Jul;35(7):2108-2113. doi: 10.1038/s41375-020-01108-x. Epub 2020 Dec 17. No abstract available. PMID 33328591
- [Background] Salles, G., Dyer, MJS,. Hodson, DJ., et-al. Updated Preliminary Results of a Phase 1b Dose Escalation and Dose Expansion Study of Tirabrutinib in Combination with Entospletinib in Patients with B-Cell Lymphoma. Blood 2018; 132 (Supplement 1): 5344.
- [Background] Walter HS, Rule SA, Dyer MJ, Karlin L, Jones C, Cazin B, Quittet P, Shah N, Hutchinson CV, Honda H, Duffy K, Birkett J, Jamieson V, Courtenay-Luck N, Yoshizawa T, Sharpe J, Ohno T, Abe S, Nishimura A, Cartron G, Morschhauser F, Fegan C, Salles G. A phase 1 clinical trial of the selective BTK inhibitor ONO/GS-4059 in relapsed and refractory mature B-cell malignancies. Blood. 2016 Jan 28;127(4):411-9. doi: 10.1182/blood-2015-08-664086. Epub 2015 Nov 5. PMID 26542378
- [Background] Walter HS, Salles GA, Dyer MJ. New Agents to Treat Chronic Lymphocytic Leukemia. N Engl J Med. 2016 Jun 2;374(22):2185-6. doi: 10.1056/NEJMc1602674. No abstract available. PMID 27248633
- [Background] Morschhauser, F., Radford, J., Ysebaert, L., et-al. Updated Preliminary Results of a Phase 1b Dose Escalation and Dose Expansion Study of Tirabrutinib in Combination with Idelalisib in Patients with B-Cell Lymphoma. Blood 2018; 132 (Supplement 1): 5345.
- [Background] Walter HS, Jayne S, Rule SA, Cartron G, Morschhauser F, Macip S, Karlin L, Jones C, Herbaux C, Quittet P, Shah N, Hutchinson CV, Fegan C, Yang Y, Mitra S, Salles G, Dyer MJS. Long-term follow-up of patients with CLL treated with the selective Bruton's tyrosine kinase inhibitor ONO/GS-4059. Blood. 2017 May 18;129(20):2808-2810. doi: 10.1182/blood-2017-02-765115. Epub 2017 Apr 4. No abstract available. PMID 28377400
- [Derived] Yahiaoui A, Meadows SA, Sorensen RA, Cui ZH, Keegan KS, Brockett R, Chen G, Queva C, Li L, Tannheimer SL. PI3Kdelta inhibitor idelalisib in combination with BTK inhibitor ONO/GS-4059 in diffuse large B cell lymphoma with acquired resistance to PI3Kdelta and BTK inhibitors. PLoS One. 2017 Feb 8;12(2):e0171221. doi: 10.1371/journal.pone.0171221. eCollection 2017. PMID 28178345
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-401-1757

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in France, the United Kingdom and the United States.
Pre-assignment Details: 248 participants were screened. 203 participants were enrolled, 197 participants were enrolled to receive treatment in Combinations I to IV and Group V. 5 participants rolled over from another tirabrutinib study (GS-US-401-1787) and 1 from this study (GS-US-401-1757) was re-assigned to Group VI to continue with tirabrutinib and be monitored for long-term safety. Per pre-specified analysis, participants in Group VI were analyzed based on the disease type.
Groups:
- Combination I (Tirabrutinib 20 mg QD+ Idelalisib 50 mg BID): Participants received tirabrutinib 20 mg tablet once daily (QD) for up to 209 weeks and idelalisib 50 mg tablet twice daily (BID) orally for up to 120 weeks. Both drugs were administered for 28-day cycles.
- Combination I (Tirabrutinib 40 mg QD+ Idelalisib 50 mg BID): Participants received tirabrutinib 40 mg tablet QD for up to 251 weeks and idelalisib 50 mg tablet BID orally, for up to 245 weeks. Both drugs were administered for 28-day cycles.
- Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID): Participants received tirabrutinib 80 mg tablet QD for up to 212 weeks and idelalisib 50 mg tablet BID orally, for up to 26 weeks. Both drugs were administered for 28-day cycles.
- Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD): Participants received tirabrutinib 80 mg tablet QD for up to 227 weeks and idelalisib 100 mg tablet QD orally, for up to 227 weeks. Both drugs were administered for 28-day cycles.
- Combination I (Tirabrutinib 160 mg QD+ Idelalisib 100 mg QD): Participants received tirabrutinib 160 mg tablet QD for up to 151 weeks and idelalisib 100 mg tablet QD orally, for up to 151 weeks. Both drugs were administered for 28-day cycles.
- Combination I (Tirabrutinib 20 mg BID+ Idelalisib 50 mg BID): Participants received tirabrutinib 20 mg tablet BID for up to 207 weeks and idelalisib 50 mg tablet BID orally, for up to 207 weeks. Both drugs were administered for 28-day cycles.
- Combination II (Tirabrutinib 40 mg QD+ Entospletinib 200 mg QD): Participants received tirabrutinib 40 mg tablet QD for up to 250 weeks and entospletinib 200 mg tablet QD orally, for up to 250 weeks. Both drugs were administered for 28-day cycles.
- Combination II (Tirabrutinib 80 mg QD+ Entospletinib 200 mg QD): Participants received tirabrutinib 80 mg tablet QD for up to 234 weeks and entospletinib 200 mg tablet QD orally, for up to 220 weeks. Both drugs were administered for 28-day cycles.
- Combination II (Tirabrutinib 150 mg QD+ Entospletinib 200 mg QD): Participants received tirabrutinib 150 mg tablet QD for up to 103 weeks and entospletinib 200 mg tablet QD orally, for up to 88 weeks. Both drugs were administered for 28-day cycles.
- Combination II (Tirabrutinib 40 mg QD+ Entospletinib 400 mg QD): Participants received tirabrutinib 40 mg tablet QD for up to 119 weeks and entospletinib 400 mg tablet QD orally, for up to 119 weeks. Both drugs were administered for 28-day cycles.
- Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD): Participants received tirabrutinib 80 mg tablet QD for up to 232 weeks and entospletinib 400 mg tablet QD orally, for up to 229 weeks. Both drugs were administered for 28-day cycles.
- Combination II (Tirabrutinib 160 mg QD+ Entospletinib 400 mg QD): Participants received tirabrutinib 160 mg tablet QD for up to 44 weeks and entospletinib 400 mg tablet QD orally, for up to 44 weeks. Both drugs were administered for 28-day cycles.
- Combination III (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD+ Obinutuzumab 1000 mg): Participants received tirabrutinib 80 mg tablet QD for up to 199 weeks; Idelalisib 100 mg tablet QD orally for up to 199 weeks, and single dose of obinutuzumab 1000 mg intravenously (IV) for up to 22 weeks. All drugs were administered for 28-day cycles.
- Combination IV(Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD+Obinutuzumab 1000 mg): Participants received tirabrutinib 80 mg tablet QD for up to 196 weeks; entospletinib 400 mg tablet QD orally for up to 196 weeks and single dose of obinutuzumab 1000 mg IV for up to 22 weeks. All drugs were administered for 28-day cycles.
- Group V Single Agent Tirabrutinib 80 mg: Participants received tirabrutinib 80 mg tablet QD orally, for each 28-day cycle up to 194 weeks.
- Group VI Single Agent Tirabrutinib: CLL: Participants with CLL who received tirabrutinib in this or previous tirabrutinib study, continued to receive tirabrutinib at the original dose (between the range of 40 - 400 mg), tablet QD, for each 28-day cycle up to 441 weeks. Participants were monitored for long-term safety of tirabrutinib this group.
- Group VI Single Agent Tirabrutinib: NHL: Participants with NHL who received tirabrutinib in this or previous tirabrutinib study, continued to receive tirabrutinib at the original dose (between the range of 60 - 480 mg), tablet QD, for each 28-day cycle up to 441 weeks. Participants were monitored for long-term safety of tirabrutinib this group.
Period: Overall Study
Arm/Group | Combination I (Tirabrutinib 20 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 40 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 160 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 20 mg BID+ Idelalisib 50 mg BID) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 150 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 160 mg QD+ Entospletinib 400 mg QD) | Combination III (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD+ Obinutuzumab 1000 mg) | Combination IV(Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD+Obinutuzumab 1000 mg) | Group V Single Agent Tirabrutinib 80 mg | Group VI Single Agent Tirabrutinib: CLL | Group VI Single Agent Tirabrutinib: NHL
Started | 3 | 8 | 4 | 25 | 9 | 5 | 3 | 6 | 3 | 3 | 78 | 8 | 6 | 7 | 29 | 3 | 3
Rollover Participants | 1 (1 participant from Combination I rolled over to Group VI CLL disease type group and continued taking tirabrutinib monotherapy.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 8 | 4 | 25 | 9 | 4 | 3 | 6 | 3 | 3 | 78 | 8 | 6 | 7 | 29 | 3 | 3
Not completed — Progressive Disease | 2 | 2 | 1 | 11 | 7 | 3 | 2 | 1 | 1 | 2 | 45 | 6 | 2 | 2 | 10 | 1 | 1
Not completed — Investigator's Discretion | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 10 | 2 | 2 | 1 | 5 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 1 | 0 | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 8 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 4 | 1 | 0 | 0 | 1 | 0 | 1 | 6 | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 2 | 0 | 1
Not completed — Transition to the MHRA's Special Scheme | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Withdrew Consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Unacceptable Toxicity | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Not completed — Intercurrent Illness | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Combination IV (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD+Obinutuzumab 1000 mg): Participants received tirabrutinib 80 mg tablet QD for up to 196 weeks; entospletinib 400 mg tablet QD orally for up to 196 weeks and single dose of obinutuzumab 1000 mg IV for up to 22 weeks. All drugs were administered for 28-day cycles.
- Group V Single Agent Tirabrutinib: Participants received tirabrutinib 80 mg tablet QD orally, for each 28-day cycle up to 194 weeks.
- Group VI Single Agent Tirabrutinib: CLL: Participants with CLL received tirabrutinib, at the original dose (20 - 160 mg), tablet QD, for each 28-day cycle up to 441 weeks.
- Group VI Single Agent Tirabrutinib: NHL: Participants with NHL received tirabrutinib, at the original dose (20 - 160 mg), tablet QD, for each 28-day cycle up to 441 weeks.
- Total: Total of all reporting groups
Arm/Group | Combination I (Tirabrutinib 20 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 40 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 160 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 20 mg BID+ Idelalisib 50 mg BID) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 150 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 160 mg QD+ Entospletinib 400 mg QD) | Combination III (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD+ Obinutuzumab 1000 mg) | Combination IV (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD+Obinutuzumab 1000 mg) | Group V Single Agent Tirabrutinib | Group VI Single Agent Tirabrutinib: CLL | Group VI Single Agent Tirabrutinib: NHL | Total
Number analyzed (Participants) | 3 | 8 | 4 | 25 | 9 | 5 | 3 | 6 | 3 | 3 | 78 | 8 | 6 | 7 | 29 | 3 | 3 | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 2 | 12 | 2 | 4 | 0 | 1 | 1 | 0 | 26 | 4 | 3 | 3 | 8 | 1 | 0 | 72
  >=65 years | 1 | 5 | 2 | 13 | 7 | 1 | 3 | 5 | 2 | 3 | 52 | 4 | 3 | 4 | 21 | 2 | 3 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (4.4) | 65 (9.7) | 62 (12.0) | 64 (13.2) | 73 (8.9) | 55 (12.8) | 70 (7.0) | 66 (11.1) | 67 (5.1) | 67 (1.2) | 68 (11.7) | 63 (11.9) | 59 (11.8) | 64 (14.4) | 70 (9.4) | 66 (4.0) | 74 (4.4) | 67 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 0 | 10 | 4 | 2 | 0 | 3 | 0 | 2 | 25 | 3 | 3 | 3 | 12 | 1 | 2 | 75
  Male | 0 | 6 | 4 | 15 | 5 | 3 | 3 | 3 | 3 | 1 | 53 | 5 | 3 | 4 | 17 | 2 | 1 | 128
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 8 | 4 | 23 | 7 | 4 | 3 | 6 | 2 | 3 | 51 | 7 | 4 | 1 | 23 | 2 | 3 | 154
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 27 | 1 | 2 | 6 | 6 | 1 | 0 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 3 | 7 | 3 | 17 | 3 | 3 | 3 | 6 | 3 | 3 | 46 | 5 | 4 | 1 | 21 | 3 | 3 | 134
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 6 | 6 | 1 | 0 | 0 | 0 | 0 | 30 | 3 | 2 | 6 | 8 | 0 | 0 | 62
Region of Enrollment [Count of Participants; unit: Participants]
  France | 0 | 2 | 2 | 8 | 6 | 1 | 1 | 0 | 1 | 2 | 35 | 7 | 4 | 7 | 7 | 0 | 0 | 83
  United Kingdom | 0 | 4 | 2 | 13 | 2 | 2 | 0 | 4 | 2 | 1 | 35 | 1 | 0 | 0 | 12 | 2 | 3 | 83
  United States | 3 | 2 | 0 | 4 | 1 | 2 | 2 | 2 | 0 | 0 | 8 | 0 | 2 | 0 | 10 | 1 | 0 | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT was defined as a ≥ Grade 3 AE that was assessed as related to study drug that occurred during the 28-day DLT assessment period with protocol-defined allowed exceptions. Any treatment-emergent adverse event (TEAE) that was, in the opinion of the Clinical Trial Steering Committee, of potential clinical significance such that further dosing exposed participants to unacceptable risk, was considered a DLT.
Time Frame: Up to 28 days
Population: The participants in the DLT Analysis Set with available data were analyzed. The DLT Analysis Set included all participants in the dose escalation, in Combination I, II, III, IV, who completed all treatment for at least 21 days within the first 28 days, or experienced a DLT prior to Day 28, inclusive.
Measure: Number; unit: percentage of participants
Arm/Group | Combination I (Tirabrutinib 20 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 40 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 160 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 20 mg BID+ Idelalisib 50 mg BID) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 150 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 160 mg QD+ Entospletinib 400 mg QD) | Combination III (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD+ Obinutuzumab 1000 mg) | Combination IV(Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD+Obinutuzumab 1000 mg)
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 4 | 5 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4
percentage of participants | 0 | 0 | 0 | 0 | 0 | 20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Objective Response Rate (ORR): Percentage of Participants With Complete Response (CR) or Partial Response (PR) at Week 12 in Participants With Non-Chronic Lymphocytic Leukemia (CLL) Type NHL
Description: ORR for Waldenstrom Macroglobulinemia(WM):CR+VGPR+PR+MPR. CR: Absence of serum monoclonal IgM protein; normal serum IgM level: complete resolution of extramedullary disease, morphologically normal bone marrow/aspirate and trephine biopsy. Very good partial response (VGPR):Detectable monoclonal IgM; ≥90% reduction in serum IgM; Complete resolution of extramedullary disease; No new signs/symptoms. PR: Monoclonal immunoglobulin M (IgM) protein is detectable ≥50% but <90% reduction in serum IgM level from baseline; reduction of extramedullary disease; no new signs or symptoms of active disease. Minor response (MPR):Detectable monoclonal IgM; ≥25% but <50% reduction in serum IgM; No progression of extramedullary disease; No new signs/symptoms. Clopper-Pearson method was used in analysis. Data is reported by disease type: WM; Follicular Lymphoma (FL);Mantle Cell Lymphoma (MCL);Small Lymphocytic Lymphoma (SLL);Marginal Zone Lymphoma (MZL);Diffuse Large B-Cell Lymphoma (DLBCL) as applicable.
Time Frame: Week 12
Population: Participants in the Full Analysis Set with non-CLL type of Non-Hodgkin's Lymphoma (NHL), were analyzed. The Full Analysis Set included all enrolled participants who took at least 1 dose of study drug. Group V did not have any participants with non-CLL type of NHL, therefore, no data is reported for this arm.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combination I (Tirabrutinib 20 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 40 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 160 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 20 mg BID+ Idelalisib 50 mg BID) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 150 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 160 mg QD+ Entospletinib 400 mg QD) | Combination III (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD+ Obinutuzumab 1000 mg) | Combination IV (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD+Obinutuzumab 1000 mg) | Group V Single Agent Tirabrutinib 80 mg
Number analyzed (Participants) | 2 | 3 | 3 | 19 | 9 | 4 | 3 | 3 | 3 | 3 | 71 | 8 | 6 | 7 | 0
percentage of participants
  Disease Subtype: FL: number analyzed (Participants) | 0 | 2 | 1 | 5 | 0 | 2 | 0 | 2 | 1 | 1 | 22 | 0 | 4 | 5 | 0
  Disease Subtype: FL |  | 0 [0 to 84.2] | 0 [0 to 97.5] | 20.0 [0.5 to 71.6] |  | 0 [0 to 84.2] |  | 50.0 [1.3 to 98.7] | 100.0 [2.5 to 100.0] | 0 [0 to 97.5] | 18.2 [5.2 to 40.3] |  | 25.0 [0.6 to 80.6] | 40.0 [5.3 to 85.3] |
  Disease Subtype: MCL: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 10 | 0 | 1 | 0 | 0
  Disease Subtype: MCL |  | 0 [0 to 97.5] |  |  |  |  | 0 [0 to 97.5] |  |  |  | 60.0 [26.2 to 87.8] |  | 100.0 [2.5 to 100.0] |  |
  Disease Subtype: SLL: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Disease Subtype: SLL | 50.0 [1.3 to 98.7] |  |  |  |  |  | 0 [0 to 84.2] |  |  |  |  |  |  |  |
  Disease Subtype: MZL: number analyzed (Participants) | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 4 | 0 | 1 | 2 | 0
  Disease Subtype: MZL |  |  | 100.0 [2.5 to 100.0] | 33.3 [0.8 to 90.6] |  | 0 [0 to 97.5] |  |  |  | 0 [0 to 97.5] | 50.0 [6.8 to 93.2] |  | 100.0 [2.5 to 100] | 50.0 [1.3 to 98.7] |
  Disease Subtype: WM: number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 1 | 7 | 0 | 0 | 0 | 0
  Disease Subtype: WM |  |  |  | 100.0 [39.8 to 100.0] |  | 0 [0 to 97.5] |  |  |  | 0 [0 to 97.5] | 42.9 [9.9 to 81.6] |  |  |  |
  Disease Subtype: DLBCL: number analyzed (Participants) | 0 | 0 | 1 | 7 | 9 | 0 | 0 | 1 | 2 | 0 | 28 | 8 | 0 | 0 | 0
  Disease Subtype: DLBCL |  |  | 0 [0 to 97.5] | 14.3 [0.4 to 57.9] | 22.2 [2.8 to 60.0] |  |  | 0 [0 to 97.5] | 100.0 [15.8 to 100.0] |  | 17.9 [6.1 to 36.9] | 12.5 [0.3 to 52.7] |  |  |

3. Primary Outcome: ORR: Percentage of Participants With CR or PR in Participants With CLL at Week 24
Description: ORR was defined as the percentage of participants who achieved a complete response (CR) or partial response (PR). CR and PR are defined in outcome measure#2. Clopper-Pearson method was used in outcome measure analysis. Percentages were rounded off.
Time Frame: Week 24
Population: Participants in the Full Analysis Set with CLL were analyzed. There were 5 arms in Combinations I and II that did not have participants with CLL type of NHL. Also, Combinations III and IV did not have any participants with CLL type of NHL, therefore, no data is reported for these arms.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Combination I (Tirabrutinib 20 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 40 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 160 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 20 mg BID+ Idelalisib 50 mg BID) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 150 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 160 mg QD+ Entospletinib 400 mg QD) | Combination III (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD+ Obinutuzumab 1000 mg) | Combination IV(Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD+Obinutuzumab 1000 mg) | Group V Single Agent Tirabrutinib 80 mg
Number analyzed (Participants) | 1 | 5 | 1 | 6 | 0 | 1 | 0 | 3 | 0 | 0 | 7 | 0 | 0 | 0 | 29
percentage of participants | 100.0 [2.5 to 100] | 80.0 [28.4 to 99.5] | 100.0 [2.5 to 100] | 66.7 [22.3 to 95.7] |  | 100.0 [2.5 to 100] |  | 66.7 [9.4 to 99.2] |  |  | 28.6 [3.7 to 71] |  |  |  | 79.3 [60.3 to 92]

4. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product or other protocol-imposed intervention, regardless of attribution. TEAEs were defined as an AE that onset in the period from the first dose of study treatment to 30 days after the last dose of study treatment. Percentages were rounded off.
Time Frame: First dose up to last dose date (up to 441 weeks) plus 30 days
Population: The Safety Analysis Set included all participants who took at least 1 dose of any study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Combination I (Tirabrutinib 20 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 40 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 160 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 20 mg BID+ Idelalisib 50 mg BID) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 150 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 160 mg QD+ Entospletinib 400 mg QD) | Combination III (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD+ Obinutuzumab 1000 mg) | Combination IV(Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD+Obinutuzumab 1000 mg) | Group V Single Agent Tirabrutinib 80 mg | Group VI Single Agent Tirabrutinib: CLL | Group VI Single Agent Tirabrutinib: NHL
Number analyzed (Participants) | 3 | 8 | 4 | 25 | 9 | 5 | 3 | 6 | 3 | 3 | 78 | 8 | 6 | 7 | 29 | 3 | 3
percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 96.2 | 75.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

5. Secondary Outcome: ORR: Percentage of Participants With Complete Response (CR) or Partial Response (PR) in the Dose Escalation and Expansion Phase
Description: ORR for WM is CR + VGPR + PR + MPR. CR, PR, VGPR and MPR are defined in outcome measure#2. Clopper-Pearson method was used in outcome measure analysis. Percentages were rounded off. Data is reported by disease type: CLL ; FL; MCL; MZL; SLL; WM; DLBCL.
Time Frame: Up to 281 weeks
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Combination IV (Tirabrutinib 80 mg QD+Entospletinib 400 mg QD+ Obinutuzumab 1000 mg): Participants received tirabrutinib 80 mg tablet QD for up to 196 weeks; entospletinib 400 mg tablet QD orally for up to 196 weeks and single dose of obinutuzumab 1000 mg IV for up to 22 weeks. All drugs were administered for 28-day cycles.
Arm/Group | Combination I (Tirabrutinib 20 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 40 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 160 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 20 mg BID+ Idelalisib 50 mg BID) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 150 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 160 mg QD+ Entospletinib 400 mg QD) | Combination III (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD+ Obinutuzumab 1000 mg) | Combination IV (Tirabrutinib 80 mg QD+Entospletinib 400 mg QD+ Obinutuzumab 1000 mg) | Group V Single Agent Tirabrutinib 80 mg
Number analyzed (Participants) | 3 | 8 | 4 | 25 | 9 | 5 | 3 | 6 | 3 | 3 | 78 | 8 | 6 | 7 | 29
percentage of participants
  Disease Subtype: CLL: number analyzed (Participants) | 1 | 5 | 1 | 6 | 0 | 1 | 0 | 3 | 0 | 0 | 7 | 0 | 0 | 0 | 29
  Disease Subtype: CLL | 100.0 [2.5 to 100.0] | 100.0 [47.8 to 100.0] | 100.0 [2.5 to 100.0] | 83.3 [35.9 to 99.6] |  | 100.0 [2.5 to 100.0] |  | 100.0 [29.2 to 100.0] |  |  | 100.0 [59 to 100.0] |  |  |  | 86.2 [68.3 to 96.1]
  Disease Subtype: FL: number analyzed (Participants) | 0 | 2 | 1 | 5 | 0 | 2 | 0 | 2 | 1 | 1 | 22 | 0 | 4 | 5 | 0
  Disease Subtype: FL |  | 0 [0 to 84.2] | 0 [0 to 97.5] | 20.0 [0.5 to 71.6] |  | 50.0 [1.3 to 98.7] |  | 50.0 [1.3 to 98.7] | 100.0 [2.5 to 100.0] | 100.0 [2.5 to 100.0] | 36.4 [17.2 to 59.3] |  | 75.0 [19.4 to 99.4] | 60.0 [14.7 to 94.7] |
  Disease Subtype: MCL: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 10 | 0 | 1 | 0 | 0
  Disease Subtype: MCL |  | 100.0 [2.5 to 100.0] |  |  |  |  | 0 [0 to 97.5] |  |  |  | 70.0 [34.8 to 93.3] |  | 100.0 [2.5 to 100.0] |  |
  Disease Subtype: MZL: number analyzed (Participants) | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 4 | 0 | 1 | 2 | 0
  Disease Subtype: MZL |  |  | 100.0 [2.5 to 100.0] | 33.3 [0.8 to 90.6] |  | 0 [0 to 97.5] |  |  |  | 0 [0 to 97.5] | 50.0 [6.8 to 93.2] |  | 100.0 [2.5 to 100.0] | 50.0 [1.3 to 98.7] |
  Disease Subtype: SLL: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Disease Subtype: SLL | 50.0 [1.3 to 98.7] |  |  |  |  |  | 100.0 [15.8 to 100.0] |  |  |  |  |  |  |  |
  Disease Subtype: WM: number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 1 | 7 | 0 | 0 | 0 | 0
  Disease Subtype: WM |  |  |  | 100.0 [39.8 to 100.0] |  | 0 [0 to 97.5] |  |  |  | 100.0 [2.5 to 100.0] | 85.7 [42.1 to 99.6] |  |  |  |
  Disease Subtype: DLBCL: number analyzed (Participants) | 0 | 0 | 1 | 7 | 9 | 0 | 0 | 1 | 2 | 0 | 28 | 8 | 0 | 0 | 0
  Disease Subtype: DLBCL |  |  | 0 [0 to 97.5] | 14.3 [0.4 to 57.9] | 33.3 [7.5 to 70.1] |  |  | 0 [0 to 97.5] | 100.0 [15.8 to 100.0] |  | 25.0 [10.7 to 44.9] | 12.5 [0.3 to 52.7] |  |  |

6. Secondary Outcome: Progression Free Survival (PFS) During the Dose Escalation Phase and Dose Expansion Phase
Description: PFS was defined as the interval from the start of the study therapy to the earlier of the first documentation of definite disease progression (PD) or death from any cause. PD: ≥ 25% increase in serum IgM level from lowest nadir (requires confirmation) and/or progression in clinical features attributable to the disease. Kaplan-Meier (KM) estimate were used in outcome measure analysis. Data is reported by disease type: CLL; FL; MCL; MZL; other NHL; DLBCL.
Time Frame: Up to 281 weeks
Population: The participants in the Full Analysis Set were analyzed. For Cohort III and IV, data for PFS was not available by disease type due to low number of participants with events. Data is reported together for all participants in Other NHL category.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination I (Tirabrutinib 20 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 40 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 160 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 20 mg BID+ Idelalisib 50 mg BID) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 150 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 160 mg QD+ Entospletinib 400 mg QD) | Combination III (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD+ Obinutuzumab 1000 mg) | Combination IV(Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD+Obinutuzumab 1000 mg) | Group V Single Agent Tirabrutinib 80 mg
Number analyzed (Participants) | 3 | 8 | 4 | 25 | 9 | 5 | 3 | 6 | 3 | 3 | 78 | 8 | 6 | 7 | 29
months
  Disease Subtype: CLL: number analyzed (Participants) | 1 | 5 | 1 | 6 | 0 | 1 | 0 | 3 | 0 | 0 | 7 | 0 | 0 | 0 | 29
  Disease Subtype: CLL | NA [NA to NA] — Median, Lower and Upper limit of Confidence interval (CI), were not estimable due to low number of participants with events. | NA [20.8 to NA] — Median and Upper limit of CI were not estimable due to low number of participants with events. | 31.8 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. | NA [8.3 to NA] — Median and Upper limit of CI were not estimable due to low number of participants with events. |  | 39.6 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. |  | NA [NA to NA] — Median, Lower and Upper limit of CI were not estimable due to low number of participants with events. |  |  | NA [NA to NA] — Median, Lower and Upper limit of CI were not estimable due to low number of participants with events. |  |  |  | NA [NA to NA] — Median, Lower and Upper limit of CI were not estimable due to low number of participants with events.
  Disease Subtype: DLBCL: number analyzed (Participants) | 0 | 0 | 1 | 7 | 9 | 0 | 0 | 1 | 2 | 0 | 28 | 8 | 0 | 0 | 0
  Disease Subtype: DLBCL |  |  | 1.4 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. | 1.5 [1.1 to 5.0] | 2.5 [1.2 to 11.0] |  |  | 1.2 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. | NA [NA to NA] — Median, Lower and Upper limit of CI were not estimable due to low number of participants with events. |  | 2.8 [1.5 to 5.3] | 2.3 [1.4 to 4.1] |  |  |
  Disease Subtype: FL: number analyzed (Participants) | 0 | 2 | 1 | 5 | 0 | 2 | 0 | 2 | 1 | 1 | 22 | 0 | 0 | 0 | 0
  Disease Subtype: FL |  | 8.2 [5.3 to 11.1] | 5.3 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. | 5.6 [1.0 to NA] — Upper limit of CI was not estimable due to low number of participants with events. |  | 12.3 [5.4 to 19.3] |  | NA [NA to NA] — Median, Lower and Upper limit of CI were not estimable due to low number of participants with events. | 19.4 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. | 19.4 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. | 11.0 [5.1 to 21.9] |  |  |  |
  Disease Subtype: MCL: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0
  Disease Subtype: MCL |  | 21.6 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. |  |  |  |  | 5.4 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. |  |  |  | 27.6 [16.8 to NA] — Upper limit of CI was not estimable due to low number of participants with events. |  |  |  |
  Disease Subtype: other NHL: number analyzed (Participants) | 2 | 0 | 1 | 7 | 0 | 2 | 2 | 0 | 0 | 2 | 11 | 0 | 6 | 7 | 0
  Disease Subtype: other NHL | 13.7 [5.5 to 21.9] |  | 6.0 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. | NA [2.5 to NA] — Median and Upper limit of CI were not estimable due to low number of participants with events. |  | 2.6 [1.2 to 4.0] | 56.9 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. |  |  | NA [6.6 to NA] — Median and Upper limit of CI were not estimable due to low number of participants with events. | NA [8.6 to NA] — Median and Upper limit of CI were not estimable due to low number of participants with events. |  | NA [5.6 to NA] — Median and Upper limit of CI were not estimable due to low number of participants with events. | NA [5.4 to NA] — Median and Upper limit of CI were not estimable due to low number of participants with events. |

7. Secondary Outcome: Duration of Response (DOR) During the Dose Escalation Phase and Dose Expansion Phase
Description: DOR was defined as the interval from the first documentation of CR or PR to the earlier of the first documentation of definite disease progression or death from any cause. CR and PR are defined in outcome measure# 2. PD is defined in outcome measure #6. KM estimates were used in outcome measure analysis. Data is reported by disease type: CLL; FL; MCL; MZL; SLL; WM; DLBCL
Time Frame: Up to 281 weeks
Population: Participants in the Full Analysis Set with ORR were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination I (Tirabrutinib 20 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 40 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 160 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 20 mg BID+ Idelalisib 50 mg BID) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 150 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 160 mg QD+ Entospletinib 400 mg QD) | Combination III (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD+ Obinutuzumab 1000 mg) | Combination IV(Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD+Obinutuzumab 1000 mg) | Group V Single Agent Tirabrutinib 80 mg
Number analyzed (Participants) | 2 | 6 | 2 | 12 | 3 | 2 | 2 | 4 | 3 | 2 | 37 | 1 | 5 | 4 | 25
months
  Disease Subtype: CLL: number analyzed (Participants) | 1 | 5 | 1 | 5 | 0 | 1 | 0 | 3 | 0 | 0 | 7 | 0 | 0 | 0 | 25
  Disease Subtype: CLL | NA [NA to NA] — Median, Lower and Upper limit of CI were not estimable due to low number of participants with events. | NA [15.2 to NA] — Median and Upper limit of CI were not estimable due to low number of participants with events. | 26.5 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. | NA [NA to NA] — Median, Lower and Upper limit of CI were not estimable due to low number of participants with events. |  | 34.1 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. |  | NA [NA to NA] — Median, Lower and Upper limit of CI were not estimable due to low number of participants with events. |  |  | NA [NA to NA] — Median, Lower and Upper limit of CI were not estimable due to low number of participants with events. |  |  |  | NA [NA to NA] — Median, Lower and Upper limit of CI were not estimable due to low number of participants with events.
  Disease Subtype: FL: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 8 | 0 | 3 | 3 | 0
  Disease Subtype: FL |  |  |  | 3.0 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. |  | 13.8 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. |  | NA [NA to NA] — Median, Lower and Upper limit of CI were not estimable due to low number of participants with events. | 16.6 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. | 6.3 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. | 17.3 [2.3 to NA] — Upper limit of CI was not estimable due to low number of participants with events. |  | NA [NA to NA] — Median, Lower and Upper limit of CI were not estimable due to low number of participants with events. | NA [4.4 to NA] — Median and Upper limit of CI were not estimable due to low number of participants with events. |
  Disease Subtype: MCL: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 1 | 0 | 0
  Disease Subtype: MCL |  | 10.7 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. |  |  |  |  |  |  |  |  | 24.9 [14.0 to NA] — Upper limit of CI was not estimable due to low number of participants with events. |  | 2.8 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. |  |
  Disease Subtype: SLL: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Disease Subtype: SLL | 19.3 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. |  |  |  |  |  | 51.4 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. |  |  |  |  |  |  |  |
  Disease Subtype: MZL: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
  Disease Subtype: MZL |  |  | 3.3 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. | 2.5 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. |  |  |  |  |  |  | NA [NA to NA] — Median, Lower and Upper limit of CI were not estimable due to low number of participants with events. |  | 8.2 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. | NA [NA to NA] — Median, Lower and Upper limit of CI were not estimable due to low number of participants with events. |
  Disease Subtype: WM: number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 0 | 0 | 0 | 0
  Disease Subtype: WM |  |  |  | NA [20.1 to NA] — Median and Upper limit of CI were not estimable due to low number of participants with events. |  |  |  |  |  | NA [NA to NA] — Median, Lower and Upper limit of CI were not estimable due to low number of participants with events. | NA [13.9 to NA] — Median and Upper limit of CI were not estimable due to low number of participants with events. |  |  |  |
  Disease Subtype: DLBCL: number analyzed (Participants) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 2 | 0 | 7 | 1 | 0 | 0 | 0
  Disease Subtype: DLBCL |  |  |  | 3.9 [NA to NA] — Lower and Upper limit of CI were not estimable due to low number of participants with events. | NA [6.4 to NA] — Median and Upper limit of CI were not estimable due to low number of participants with events. |  |  |  | NA [NA to NA] — Median, Lower and Upper limit of CI were not estimable due to low number of participants with events. |  | 8.3 [1.4 to 23.5] | NA [NA to NA] — Median, Lower and Upper limit of CI were not estimable due to low number of participants with events. |  |  |

8. Secondary Outcome: Time to Response (TTR) During the Dose Escalation Phase and Dose Expansion Phase
Description: TTR was defined as the interval from start of treatment to the first documentation of CR or PR. CR and PR are defined in outcome measure# 2. Data is reported by disease type: CLL; FL; MCL; MZL; SLL; WM; DLBCL.
Time Frame: Up to 281 weeks
Population: Participants in the Full Analysis Set with ORR were analyzed.
Measure: Median (Full Range); unit: months
Arm/Group | Combination I (Tirabrutinib 20 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 40 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 160 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 20 mg BID+ Idelalisib 50 mg BID) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 150 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 160 mg QD+ Entospletinib 400 mg QD) | Combination III (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD+ Obinutuzumab 1000 mg) | Combination IV(Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD+Obinutuzumab 1000 mg) | Group V Single Agent Tirabrutinib 80 mg
Number analyzed (Participants) | 2 | 6 | 2 | 12 | 3 | 2 | 2 | 4 | 3 | 2 | 37 | 1 | 5 | 4 | 25
months
  Disease Subtype: CLL: number analyzed (Participants) | 1 | 5 | 1 | 5 | 0 | 1 | 0 | 3 | 0 | 0 | 7 | 0 | 0 | 0 | 25
  Disease Subtype: CLL | 2.7 [2.7 to 2.7] | 5.6 [5.4 to 5.8] | 5.4 [5.4 to 5.4] | 5.6 [4.6 to 8.0] |  | 5.6 [5.6 to 5.6] |  | 5.4 [4.4 to 5.9] |  |  | 5.9 [5.4 to 6.8] |  |  |  | 5.5 [2.7 to 5.9]
  Disease Subtype: FL: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 8 | 0 | 3 | 3 | 0
  Disease Subtype: FL |  |  |  | 2.6 [2.6 to 2.6] |  | 5.5 [5.5 to 5.5] |  | 2.8 [2.8 to 2.8] | 2.8 [2.8 to 2.8] | 13.0 [13.0 to 13.0] | 3.7 [2.8 to 11.0] |  | 3.9 [2.6 to 9.2] | 2.9 [2.6 to 4.6] |
  Disease Subtype: MCL: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 1 | 0 | 0
  Disease Subtype: MCL |  | 10.8 [10.8 to 10.8] |  |  |  |  |  |  |  |  | 2.8 [2.8 to 8.4] |  | 2.8 [2.8 to 2.8] |  |
  Disease Subtype: SLL: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Disease Subtype: SLL | 2.7 [2.7 to 2.7] |  |  |  |  |  | 5.5 [5.4 to 5.6] |  |  |  |  |  |  |  |
  Disease Subtype: MZL: number analyzed (Participants) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
  Disease Subtype: MZL |  |  | 2.8 [2.8 to 2.8] | 2.9 [2.9 to 2.9] |  |  |  |  |  |  | 2.7 [2.7 to 2.8] |  | 2.7 [2.7 to 2.7] | 2.8 [2.8 to 2.8] |
  Disease Subtype: WM: number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 0 | 0 | 0 | 0
  Disease Subtype: WM |  |  |  | 2.8 [2.6 to 3.0] |  |  |  |  |  | 17.5 [17.5 to 17.5] | 4.1 [2.8 to 9.1] |  |  |  |
  Disease Subtype: DLBCL: number analyzed (Participants) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 2 | 0 | 7 | 1 | 0 | 0 | 0
  Disease Subtype: DLBCL |  |  |  | 1.6 [1.6 to 1.6] | 1.8 [1.4 to 4.6] |  |  |  | 1.9 [1.1 to 2.8] |  | 1.5 [1.3 to 13.0] | 1.6 [1.6 to 1.6] |  |  |

9. Secondary Outcome: Percentage of Participants Who Achieved Minimal Residual Negative Disease (< 1 Leukemia Cell/10,000 Leukocytes) During the Dose Escalation Phase and Dose Expansion Phase in Participants With CLL
Description: Achieving Minimal Residual Disease was defined as < 1 leukemia cell/10,000 leukocytes (10-4) in participants who have also achieved a CR. CR is defined in outcome measure #2.
Time Frame: Up to 281 weeks
Population: Participants in the All Enrolled Analysis Set with CLL were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Combination I (Tirabrutinib 20 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 40 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 160 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 20 mg BID+ Idelalisib 50 mg BID) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 150 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 160 mg QD+ Entospletinib 400 mg QD) | Combination III (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD+ Obinutuzumab 1000 mg) | Combination IV(Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD+Obinutuzumab 1000 mg) | Group V Single Agent Tirabrutinib 80 mg
Number analyzed (Participants) | 1 | 5 | 1 | 6 | 0 | 1 | 0 | 3 | 0 | 0 | 7 | 0 | 0 | 0 | 29
percentage of participants | 0 | 40 | 0 | 16.7 |  | 0 |  | 0 |  |  | 28.6 |  |  |  | 20.7

10. Secondary Outcome: Pharmacokinetic (PK) Parameter: AUCtau of Tirabrutinib 80 mg
Description: AUCtau was defined as concentration of drug over time. Area under the concentration verses time curve over the dosing interval (AUctau). The data for AUCtau is reported for tirabrutinib 80 mg as monotherapy and in combination with idelalisib 50 mg and 100 mg and entospletinib 200 mg and 400 mg.
Time Frame: Cycle 1 Day 8: Predose and 0.5, 1, 2, 3, 4, 6, 8 and 24 hours postdose
Population: Participants in the tirabrutinib PK Analysis Set with available data were analyzed. The PK Analysis Set included participants who received at least 1 dose of study drug and had at least 1 non-missing post-dose concentration value reported by the PK laboratory.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD): Participants received tirabrutinib 40 mg tablet QD for up to 119 weeks and entospletinib 400 mg tablet QD orally, for up to 119 weeks. Both drugs were administered for 28-day cycles.
Arm/Group | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD) | Group V Single Agent Tirabrutinib
Number analyzed (Participants) | 4 | 2 | 3 | 3 | 9
ng*h/mL | 984.0 (342.18) | 1205.6 (245.89) | 1794.1 (181.15) | 1251.6 (387.46) | 1088.8 (545.52)

11. Secondary Outcome: PK Parameter: Cmax of Tirabrutinib 80 mg
Description: Cmax was defined as the maximum observed concentration of drug. The data for Cmax is reported for tirabrutinib 80 mg as monotherapy and in combination with idelalisib 50 mg and 100 mg and entospletinib 200 mg and 400 mg.
Time Frame: Cycle 1 Day 8: Predose and 0.5, 1, 2, 3, 4, 6, 8 and 24 hours postdose
Population: The participants in the tirabrutinib PK analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD) | Group V Single Agent Tirabrutinib
Number analyzed (Participants) | 4 | 2 | 3 | 3 | 10
ng/mL | 192.3 (58.21) | 219.5 (12.02) | 304.7 (34.67) | 246.3 (11.37) | 215.2 (66.10)

12. Secondary Outcome: PK Parameter: AUCtau of Idelalisib When Given in Combination With Tirabrutinib
Description: AUCtau was defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Time Frame: Cycle 1 Day 8: Predose and 0.5, 1, 2, 3, 4, 6, 8 and 24 hours postdose
Population: Participants in the Idelalisib PK analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Combination I (Tirabrutinib 20 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 40 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 160 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 20 mg BID+ Idelalisib 50 mg BID)
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 4 | 5
h*ng/mL | 6620.6 (661.19) | 5433.2 (1287.95) | 6735.0 (1859.79) | 9488.0 (3263.44) | 19305.4 (5616.53) | 7093.0 (4025.04)

13. Secondary Outcome: PK Parameter: Cmax of Idelalisib When Given in Combination With Tirabrutinib
Description: Cmax was defined as the maximum observed concentration of drug.
Time Frame: Cycle 1 Day 8: Predose and 0.5, 1, 2, 3, 4, 6, 8 and 24 hours postdose
Population: Participants in the Idelalisib PK analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Combination I (Tirabrutinib 20 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 40 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 160 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 20 mg BID+ Idelalisib 50 mg BID)
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 4 | 5
ng/mL | 1920.0 (252.39) | 1893.3 (750.82) | 1324.8 (389.65) | 1790.0 (268.70) | 3325.0 (481.28) | 1844.0 (518.58)

14. Secondary Outcome: PK Parameter: AUCtau of Metabolite of Idelalisib (GS-563117) When Given in Combination With Tirabrutinib
Description: as for outcome 12
Time Frame: Cycle 1 Day 8: Predose and 0.5, 1, 2, 3, 4, 6, 8 and 24 hours postdose
Population: Participants in the Idelalisib Metabolite PK Analysis Set with available data were analyzed. The Idelalisib Metabolite PK Analysis Set included participants who received at least 1 dose of study drug and had at least 1 nonmissing post-dose concentration value reported by the PK laboratory.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Combination I (Tirabrutinib 20 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 40 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 160 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 20 mg BID+ Idelalisib 50 mg BID)
Number analyzed (Participants) | 3 | 3 | 2 | 2 | 3 | 3
h*ng/mL | 19922.6 (9354.47) | 22519.6 (8233.77) | 41327.5 (20049.44) | 49192.7 (15719.52) | 36824.3 (9670.67) | 225371.5 (22931.89)

15. Secondary Outcome: PK Parameter: Cmax of Metabolite of Idelalisib (GS-563117) When Given in Combination With Tirabrutinib
Description: Cmax was defined as the maximum observed concentration of drug.
Time Frame: Cycle 1 Day 8: Predose and 0.5, 1, 2, 3, 4, 6, 8 and 24 hours postdose
Population: Participants in the Idelalisib Metabolite PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Combination I (Tirabrutinib 20 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 40 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 160 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 20 mg BID+ Idelalisib 50 mg BID)
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 4 | 5
ng/mL | 2723.3 (1045.10) | 2760.0 (1105.31) | 2542.5 (1820.54) | 3415.0 (360.62) | 2592.5 (503.48) | 3682.0 (1950.35)

16. Secondary Outcome: PK Parameter: AUCtau of Entospletinib When Given in Combination With Tirabrutinib
Description: as for outcome 12
Time Frame: Cycle 1 Day 8: Predose and 0.5, 1, 2, 3, 4, 6, 8 and 24 hours postdose
Population: Participants in the Entospletinib PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 150 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 160 mg QD+ Entospletinib 400 mg QD)
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 3 | 4
h*ng/mL | 7738.7 (1793.68) | 4266.2 (1574.30) | 9968.3 (295.69) | 14027.8 (6979.18) | 12959.9 (2250.66) | 6196.8 (1018.98)

17. Secondary Outcome: PK Parameter: Cmax of Entospletinib When Given in Combination With Tirabrutinib
Description: Cmax was defined as the maximum observed concentration of drug.
Time Frame: Cycle 1 Day 8: Predose and 0.5, 1, 2, 3, 4, 6, 8 and 24 hours postdose
Population: Participants in the Entospletinib PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 150 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 160 mg QD+ Entospletinib 400 mg QD)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 4
ng/mL | 876.0 (367.98) | 707.7 (397.04) | 697.0 (313.93) | 1498.7 (619.57) | 1330.7 (382.0) | 861.0 (276.17)

ADVERSE EVENTS:
Time Frame: Up to 441 weeks plus 30 days
Description: All-Cause mortality: All Enrolled Analysis Set includes all participants who received a participant ID number in the study after screening.
  Adverse events: The Safety Analysis Set included all participants who took at least 1 dose of any study treatment, with treatment assignment designated according to the actual treatment received.
Arm/Group | Combination I (Tirabrutinib 20 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 40 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 160 mg QD+ Idelalisib 100 mg QD) | Combination I (Tirabrutinib 20 mg BID+ Idelalisib 50 mg BID) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 150 mg QD+ Entospletinib 200 mg QD) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD) | Combination II (Tirabrutinib 160 mg QD+ Entospletinib 400 mg QD) | Combination III (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD+ Obinutuzumab 1000 mg) | Combination IV(Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD+Obinutuzumab 1000 mg) | Group V Single Agent Tirabrutinib 80 mg | Group VI Single Agent Tirabrutinib: CLL | Group VI Single Agent Tirabrutinib: NHL
All-Cause Mortality (participants affected / at risk) | 0/3 | 2/8 | 1/4 | 6/25 | 1/9 | 2/5 | 0/3 | 0/6 | 0/3 | 0/3 | 8/78 | 2/8 | 1/6 | 1/7 | 3/29 | 0/3 | 1/3
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/8 | 2/4 | 13/25 | 2/9 | 4/5 | 3/3 | 4/6 | 1/3 | 1/3 | 36/78 | 2/8 | 4/6 | 7/7 | 10/29 | 1/3 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 8/8 | 4/4 | 24/25 | 9/9 | 5/5 | 3/3 | 6/6 | 3/3 | 3/3 | 73/78 | 5/8 | 6/6 | 7/7 | 29/29 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination I (Tirabrutinib 20 mg QD+ Idelalisib 50 mg BID) (N=3) | Combination I (Tirabrutinib 40 mg QD+ Idelalisib 50 mg BID) (N=8) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID) (N=4) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD) (N=25) | Combination I (Tirabrutinib 160 mg QD+ Idelalisib 100 mg QD) (N=9) | Combination I (Tirabrutinib 20 mg BID+ Idelalisib 50 mg BID) (N=5) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 200 mg QD) (N=3) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 200 mg QD) (N=6) | Combination II (Tirabrutinib 150 mg QD+ Entospletinib 200 mg QD) (N=3) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 400 mg QD) (N=3) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD) (N=78) | Combination II (Tirabrutinib 160 mg QD+ Entospletinib 400 mg QD) (N=8) | Combination III (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD+ Obinutuzumab 1000 mg) (N=6) | Combination IV(Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD+Obinutuzumab 1000 mg) (N=7) | Group V Single Agent Tirabrutinib 80 mg (N=29) | Group VI Single Agent Tirabrutinib: CLL (N=3) | Group VI Single Agent Tirabrutinib: NHL (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Death, not otherwise specified (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Cytokine storm (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspergillus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Covid-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster disseminated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral discitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Norovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural fever (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biphasic mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bladder transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vasculitic ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination I (Tirabrutinib 20 mg QD+ Idelalisib 50 mg BID) (N=3) | Combination I (Tirabrutinib 40 mg QD+ Idelalisib 50 mg BID) (N=8) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 50 mg BID) (N=4) | Combination I (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD) (N=25) | Combination I (Tirabrutinib 160 mg QD+ Idelalisib 100 mg QD) (N=9) | Combination I (Tirabrutinib 20 mg BID+ Idelalisib 50 mg BID) (N=5) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 200 mg QD) (N=3) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 200 mg QD) (N=6) | Combination II (Tirabrutinib 150 mg QD+ Entospletinib 200 mg QD) (N=3) | Combination II (Tirabrutinib 40 mg QD+ Entospletinib 400 mg QD) (N=3) | Combination II (Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD) (N=78) | Combination II (Tirabrutinib 160 mg QD+ Entospletinib 400 mg QD) (N=8) | Combination III (Tirabrutinib 80 mg QD+ Idelalisib 100 mg QD+ Obinutuzumab 1000 mg) (N=6) | Combination IV(Tirabrutinib 80 mg QD+ Entospletinib 400 mg QD+Obinutuzumab 1000 mg) (N=7) | Group V Single Agent Tirabrutinib 80 mg (N=29) | Group VI Single Agent Tirabrutinib: CLL (N=3) | Group VI Single Agent Tirabrutinib: NHL (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 2 | 0 | 0 | 8 | 0 | 1 | 2 | 5 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 2 | 8 | 1 | 2 | 1 | 3 | 0 | 1 | 14 | 0 | 2 | 4 | 4 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 4 | 3 | 1 | 0 | 0 | 0 | 0 | 8 | 0 | 1 | 3 | 2 | 1 | 0
Warm autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Gilbert's syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Porokeratosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Macular degeneration (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Macular hole (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scleritis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Xerophthalmia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 3 | 1 | 0 | 0 | 2 | 0 | 0 | 9 | 2 | 1 | 2 | 3 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Apical granuloma (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breath odour (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 1 | 3 | 1 | 4 | 0 | 2 | 0 | 1 | 11 | 0 | 2 | 3 | 8 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 5 | 1 | 5 | 4 | 2 | 0 | 3 | 1 | 0 | 24 | 3 | 3 | 2 | 10 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 0 | 2 | 2 | 1 | 1 | 1 | 1 | 1 | 9 | 0 | 1 | 0 | 4 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 5 | 1 | 0 | 0 | 1 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Lip disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth swelling (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 1 | 3 | 1 | 2 | 0 | 1 | 0 | 0 | 18 | 1 | 2 | 1 | 10 | 0 | 0
Oral blood blister (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 1 | 2 | 0 | 2 | 0 | 0 | 11 | 1 | 1 | 0 | 2 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 3 | 0 | 1 | 1 | 0 | 0 | 1 | 17 | 2 | 1 | 3 | 3 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Cyst (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 3 | 1 | 2 | 1 | 4 | 2 | 0 | 21 | 0 | 1 | 1 | 8 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperthermia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Oedema peripheral (General disorders) | 2 | 0 | 1 | 3 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 6 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 0 | 2 | 0 | 0
Peripheral swelling (General disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 3 | 2 | 1 | 3 | 1 | 1 | 0 | 2 | 0 | 1 | 14 | 0 | 1 | 1 | 3 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bartholinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 2 | 2 | 5 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cholangitis infective (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 5 | 0 | 1 | 0 | 6 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemophilus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Infected bite (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Infected cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 7 | 0 | 2 | 1 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 6 | 0 | 0 | 0 | 5 | 2 | 0
Lymph gland infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 4 | 0 | 2 | 0 | 2 | 0 | 0 | 13 | 0 | 1 | 3 | 4 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Oral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 5 | 0 | 0 | 0 | 5 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 2 | 2 | 5 | 0 | 0 | 0 | 2 | 1 | 0 | 9 | 0 | 1 | 2 | 5 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 0 | 1 | 0 | 3 | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tongue fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Toxocariasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 4 | 1 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 6 | 0 | 1 | 0 | 7 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 5 | 0 | 1 | 0 | 3 | 1 | 1
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Vulvitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 2 | 0 | 4 | 0 | 1 | 0 | 2 | 0 | 1 | 15 | 0 | 0 | 0 | 6 | 0 | 0
Eye abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 8 | 0 | 0 | 0 | 3 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 7 | 1 | 1 | 0 | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 6 | 1 | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0
Blood urine present (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Influenza A virus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sars-cov-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 4 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3 | 0 | 3 | 0 | 0 | 0 | 0 | 9 | 0 | 1 | 1 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 6 | 1 | 1 | 0 | 1 | 0 | 0 | 13 | 0 | 2 | 1 | 6 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 4 | 1 | 2 | 0 | 3 | 0 | 1 | 14 | 1 | 1 | 0 | 6 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 2 | 0 | 4 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 4 | 0 | 1 | 0 | 2 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neurofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Akathisia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 9 | 0 | 1 | 2 | 7 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 2 | 2 | 2 | 0 | 1 | 0 | 0 | 9 | 0 | 1 | 0 | 4 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 3 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mixed anxiety and depressive disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast induration (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pelvic organ prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 4 | 2 | 2 | 0 | 3 | 1 | 0 | 14 | 0 | 4 | 2 | 7 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 4 | 1 | 2 | 0 | 1 | 0 | 1 | 12 | 0 | 2 | 0 | 4 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 7 | 0 | 0 | 0 | 3 | 0 | 0
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 5 | 0 | 0 | 0 | 6 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 12 | 0 | 1 | 1 | 4 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 11 | 1 | 2 | 1 | 2 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 1 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 7 | 1 | 1 | 0 | 2 | 1 | 0 | 11 | 1 | 1 | 1 | 5 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 6 | 0 | 2 | 1 | 3 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Solar lentigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 2 | 3 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 4 | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT02457598/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT02457598/SAP_001.pdf